CLINICAL TRIAL: NCT05944562
Title: Phase I Study With an Expansion Cohort of Tulmimetostat (DZR123) in Patients With Mycosis Fungoides and Sézary Syndrome
Brief Title: Tulmimetostat (DZR123) in Patients With Mycosis Fungoides and Sézary Syndrome
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis (Industry); The Foundation for Barnes-Jewish Hospital (Other); Swim Across America (Other); Daniel E. Corbin Jr. Lymphoma Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202310037
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mycosis Fungoides; Sezary Syndrome; Mycosis Fungoides/Sezary Syndrome
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose De-Escalation Cohort: Tulmimetostat (DZR123) (Experimental): Daily DZR123 by mouth for days 1-28 of each 28-day cycle. Dose will depend on dose level assignment of 300 mg daily, 250 mg daily, or 200 mg daily.
- Dose Expansion Cohort: Tulmimetostat (DZR123) - 300 mg (Experimental): Daily DZR123by mouth for days 1-28 of each 28-day cycle. Dose will be the maximum-tolerated dose found during the dose de-escalation cohort which was 300 mg.
- Dose Expansion Cohort: Tulmimetostat (DZR123) - 200 mg (Experimental): Daily DZR123 by mouth for days 1-28 of each 28-day cycle. Dose will be 200 mg as the maximum tolerated dose of 300 mg found during the initial dose expansion cohort caused numerous dose reductions.

INTERVENTIONS:
Drug: Tulmimetostat — Patients should take DZR123 at approximately the same time every morning in a fasted state (no food for 2 hours prior and 1 hour following DZR123 dosing). Each dose of DZR123 should be taken with a glass of water and consumed over as short a time as possible.
  Other Names: DZR123

SUMMARY:
The hypotheses of this study are that single agent DZR123 will be safe and well tolerated in patients with advanced (stage IB-IVB) mycosis fungoides (MF)/Sézary syndrome (SS) who have had at least one prior systemic therapy, and that in these patients, DZR123 will demonstrate efficacy and be worth of further study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed mycosis fungoides or Sézary syndrome, stages IB to IVB with measurable disease and/or detectable blood involvement based on the Global Response Criteria for CTCL (Olsen et al., 2022).
* Received at least one prior line of systemic therapy.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Adequate counts and organ function as defined below:

  * ANC ≥ 0.7 x 109/L, without growth factor support (filgrastim or pegfilgrastim) for at least 14 days
  * Platelets ≥ 75 x 109/L, without platelet transfusion for at least 14 days
  * Hemoglobin ≥ 8.0 g/dL, with or without transfusion
  * Serum total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault (using actual body weight) for patients with creatinine levels above institutional normal OR serum creatinine ≤ 1.5 x ULN
* Patients with treated brain metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no evidence of progression.
* The effects of DZR123 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use highly effective methods of contraception for the duration of study participation and for 183 days after the last dose of DZR123 for female patients and female partners of male patients, or for 93 days after the last dose of DZR123 for male patients and male partners of female patients. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Prior treatment with an EZH2 inhibitor.
* Patients with CNS lymmphoma.
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

  * Those with local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, high grade superficial bladder cancer and carcinoma in situ, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for ≥ 1 year prior to registration, asymptomatic breast cancer on adjuvant hormonal therapy diagnosed more than 2 years ago, adequately treated Stage 1 or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for ≥ 3 years are eligible.
* Currently receiving any other investigational agents. Concomitant use of another systemic therapy for MF/SS. Patients must have the following minimum wash-out from previous treatments:

  * At least 8 weeks for low-dose (12 Gy or less) total skin electron beam therapy (TSEBT)
  * At least 4 weeks for systemic cytotoxic anticancer agents or for tumor-targeting monoclonal antibodies (mAbs), with the exception of alemtuzumab, for which the washout is at least 16 weeks
  * At least 2 weeks or 5 half-lives for systemic retinoids, interferons, vorinostat, romidepsin, and denileukin diftitox, or anticancer investigational agents that are not defined as immunotherapy,
  * At least 2 weeks for local radiation therapy
  * At least 1 week for topical retinoids, nitrogen mustard, or imiquimod
* Taking concomitant medication(s) or food or beverage that are strong CYP3A inducers or inhibitors within 7 days prior to the first dose of study drug.
* History of allogeneic HCT within 90 days prior to the first dose of study drug.
* Clinically significant graft-versus-host disease (GVHD) or GVHD requiring systemic immunosuppressive prophylaxis or treatment.
* Previous solid organ transplant.
* Clinically significant cardiovascular disease including:

  * Myocardial infarction/stroke within 3 months prior to Day 1 of treatment
  * Unstable angina within 3 months prior to Day 1 of treatment
  * Congestive heart failure or cardiomyopathy with NYHA Class 3 or 4
  * History of clinically significant ventricular arrhythmias (e.g. ventricular tachycardia, ventricular fibrillation, Torsades de pointes)
  * Uncontrolled hypertension (as defined per institutional standards) despite 2 concomitant antihypertensive therapies
  * QT interval corrected by the Fridericia correction formula (QTcF) ≥ 480 msec at time of screening
* Major surgery within 4 weeks before starting study drug or not recovered from any effects of prior major surgery (uncomplicated central line placement or fine needle aspiration are not considered major surgery).
* Gastrointestinal disorders, i.e., ulcerative colitis, malabsorption syndrome, refractory nausea and vomiting, biliary shunt, significant bowel resection or any other condition that may significantly interfere with absorption of the study medication by the investigator's assessment.
* Uncontrolled active infection requiring IV antibiotic, antiviral, or antifungal medications within 14 days before the first dose of study drug. Infections (e.g., urinary tract infection) controlled on concurrent antimicrobial agents and antimicrobial prophylaxis per institutional guidelines are acceptable.
* Current known active or chronic infection with HIV, hepatitis B, or hepatitis C. All patients will require serologic testing to be performed within 6 months prior to C1D1.

  * Patients with chronic HBV or HCV are defined as patients with positive hepatitis B serology: Patients with a negative HBsAg and a positive HBcAb require an undetectable/negative hepatitis B DNA test (e.g. polymerase chain reaction [PCR] test) to be enrolled, and will require prophylactic antiviral treatment initiated prior to the first dose of study drug, and continued until approximately 6 to 12 months after completion of study drug(s).
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of study drug administration. Inhaled or topical steroids, steroids for physiologic or adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption) and use of these agents does not require a washout period. Topical steroids or intralesional steroids for cutaneous manifestations of MF/SS are permitted as well. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted. Patients prescribed prednisone 10 mg PO daily or less (or equivalent) will not be excluded.
* Ongoing treatment with other immunosuppressive agent including, but not limited to, methotrexate, azathioprine, anti-TNF agents, etc. with the exception of steroids.
* Clinically active or symptomatic chronic liver disease.
* Unstable or severe uncontrolled medical condition or any important medical or psychiatric illness or abnormal laboratory finding that would, in the investigator's judgment, increase the risk to the patient associated with his/her participation in this study.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 72 hours prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and grades of treatment-emergent adverse events (TEAE) | From start of treatment through 30 days after completion of treatment (estimated to be 13 months)
Rate of treatment discontinuation due to treatment-emergent adverse events (TEAE) | From start of treatment through 30 days after completion of treatment (estimated to be 13 months)

SECONDARY OUTCOMES:
Recommended phase II dose/maximum tolerated dose of CPI-0209 | Through completion of cycle 1 (28 days) of all dose de-escalation patients enrolled (each patient followed for 28 days)
  The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity (DLT) during the first cycle. In the absence of excess toxicity, the maximum tolerated dose will become the recommended phase II dose (RP2D).
Overall response rate (ORR) | At 4 months
  * Assessed according to the Global Response Criteria for CTCL.
  * Defined as the proportion of patients who achieve a partial response (PR) or complete response (CR) as measured at four months from the start of treatment
Time to maximum response | Through completion of treatment (estimated to be 12 months)
  * Assessed according to the Global Response Criteria for CTCL.
  * Quantified as the time elapsed between the date when the patient started taking CPI-0209 to the date they achieved their best overall response.
Best overall response rate | Through completion of treatment (estimated to be 12 months)
  * Assessed according to the Global Response Criteria for CTCL.
  * Defined as the total number of patients that achieve a PR or CR at any time during the study period divided by the total number of patients included in the efficacy evaluation.
Complete remission rate | Through completion of follow-up (estimated to be 36 months)
  * Assessed according to the Global Response Criteria for CTCL.
  * Defined as the total number of patients that achieve a PR or CR at any time during the study period divided by the total number of patients included in the efficacy evaluation.
Duration of response among responding patients | Through completion of follow-up (estimated to be 36 months)
  * Assessed according to the Global Response Criteria for CTCL.
  * Defined as the time elapsed between the date a patient first achieves a partial response (PR) or complete response (CR) to the date they are determined to have relapse or progression of their disease. Patients who do not achieve a PR or CR with CPI-0209 will be excluded from the duration of response analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Mehta-Shah, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu